CLINICAL TRIAL: NCT06749288
Title: Radicle Revive™ 24: A Randomized, Double-Blind, Placebo-Controlled, Direct-to-Consumer Trial Assessing the Impact of Health and Wellness Products on Hormonal Health and Associated Health Outcomes in Women With Menopausal Health Issues
Brief Title: Radicle Revive 24: A Study of Health and Wellness Products on Menopausal Health and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2414
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Menopause; Sleep Disturbance; Anxiety; Depression; Cognitive Function; Fatigue; Libido
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Intervention Model Description: Participants will be stratified then randomized to one of the study arms. Each participant will have an equal chance of being assigned to each study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control 4.1.0 (Placebo Comparator): Revive product form 4.1 - control
  Interventions: Dietary Supplement: Radicle Revive Placebo Control Form 4.1
- Active product 4.1.1 (Experimental): Revive product form 4.1 - active product 1
  Interventions: Dietary Supplement: Radicle Revive Active Study Product 4.1 Usage

INTERVENTIONS:
Dietary Supplement: Radicle Revive Placebo Control Form 4.1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo control 4.1.0
Dietary Supplement: Radicle Revive Active Study Product 4.1 Usage — Participants will use their Radicle Revive Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active product 4.1.1

SUMMARY:
A randomized, double-blind, placebo-controlled, direct-to-consumer trial assessing the impact of health and wellness products on hormonal health and associated health outcomes in women with menopausal health issues

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants (1) are females, (2) have menopausal health issues for 3 months or longer, (3) have the opportunity to improve by at least 30%, and (4) express acceptance in taking study products and not knowing the formulation identities until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and women who are pregnant or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses less pain as a primary desire
* Selects pain and/or looking to improve their pain as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* The calculated validated health survey (PRO) score during enrollment represents less than mild severity
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in a clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy or immunotherapy
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied, or a substantial safety risk: Anticoagulants, a medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, or MAO

Ages: 21 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 8A (scale 8-40; with higher scores corresponding to more severe anxiety)
Change in feelings of depression | 6 weeks
  Mean difference in depression score as assessed by PROMIS Depression 4A (scale 4-20; with higher scores corresponding to more severe depression)
Change in cognitive function | 6 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognitive Function 4A (scale 4-20; with lower scores corresponding to better cognitive function)
Change in cognitive function | 6 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; with lower scores corresponding to better cognitive function)
Change in sleep disturbance | 6 weeks
  Mean difference in sleep disturbance score as assessed by PROMIS Sleep Disturbance 4A (scale 4-20; with higher scores corresponding to more severe sleep disturbance)
Change in sleep disturbance | 6 weeks
  Mean difference in sleep disturbance score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; with higher scores corresponding to more severe sleep disturbance)
Change in fatigue | 6 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; with higher scores corresponding to more severe fatigue)
Change in feelings of depression | 6 weeks
  Mean difference in depression score as assessed by PROMIS Depression 8A (scale 8-40; with higher scores corresponding to more severe depression)
Change in fatigue | 6 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 8A (scale 8-40; with higher scores corresponding to more severe fatigue)
Change in Pain Interference | 6 weeks
  Mean difference in pain interference score as assessed by PROMIS Pain Interference 6A (scale 6-30; with higher scores corresponding to more severe pain interference)
Change in pain intensity | 6 weeks
  Mean difference in pain intensity score as assessed by PROMIS Pain Intensity 3A (scale 3-15; with higher scores corresponding to more severe pain intensity)
Change in interest in sexual activity | 6 weeks
  Mean difference in interest in sexual activity score as assessed by PROMIS Sexual Function and Satisfaction v2.0 (scale 2-10; with lower scores corresponding to less interest in sexual activity)

SECONDARY OUTCOMES:
Change in other menopausal health issues | 6 weeks
  Other menopausal health issues assessed by Radicle General Menopausal Health Issues (Point range: 10 - 48; where higher is more severe menopausal health issues)
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of achieving a MCID in anxiety, as measured by PROMIS Anxiety 4a (4-20; where lower scores indicate less anxiety).
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of achieving a MCID in anxiety, as measured by PROMIS Anxiety 8a (8-40; where lower scores indicate less anxiety).
Minimal clinically important difference (MCID) in feelings of depression | 6 weeks
  Likelihood of achieving a MCID in depression , as measured by PROMIS Depression 4a (4-20; where lower scores indicate less depression).
Minimal clinically important difference (MCID) in feelings of depression | 6 weeks
  Likelihood of achieving a MCID in depression , as measured by PROMIS Depression 8a (8-40; where lower scores indicate less depression).
Minimal clinically important difference (MCID) in cognitive function | 6 weeks
  Likelihood of achieving a MCID in cognitive function , as measured by PROMIS cognitive function 4a (4-20; where lower scores indicate poorer cognitive function).
Minimal clinically important difference (MCID) in cognitive function | 6 weeks
  Likelihood of achieving a MCID in cognitive function , as measured by PROMIS cognitive function 8a (8-40; where lower scores indicate poorer cognitive function).
Minimal clinically important difference (MCID) in sleep disturbance | 6 weeks
  Likelihood of achieving a MCID in sleep disturbance , as measured by PROMIS Sleep Disturbance 4a (4-20; where lower scores indicate less sleep disturbance).
Minimal clinically important difference (MCID) in sleep disturbance | 6 weeks
  Likelihood of achieving a MCID in sleep disturbance , as measured by PROMIS Sleep Disturbance 8a (8-40; where lower scores indicate less sleep disturbance).
Minimal clinically important difference (MCID) in fatigue | 6 weeks
  Likelihood of achieving a MCID in fatigue, as measured by PROMIS Fatigue 4a (4-20; where lower scores indicate less fatigue).
Minimal clinically important difference (MCID) in fatigue | 6 weeks
  Likelihood of achieving a MCID in fatigue, as measured by PROMIS Fatigue 8a (8-40; where lower scores indicate less fatigue).
Minimal clinically important difference (MCID) in pain interference | 6 weeks
  Likelihood of achieving a MCID in pain interference, as measured by PROMIS Pain interference (6-30; where lower scores indicate less pain interference).
Minimal clinically important difference (MCID) in pain intensity | 6 weeks
  Likelihood of achieving a MCID in pain intensity, as measured by PROMIS Pain intensity (3-15; where lower scores indicate less pain intensity).
Minimal clinically important difference (MCID) in interest in sexual function | 6 weeks
  Likelihood of achieving a MCID in interest in sexual activity, as measured by PROMIS Sexual Function and Satisfaction v2.0 (scale 2-10; with lower scores corresponding to less interest in sexual activity)

CONTACTS AND LOCATIONS:
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — http://radiclescience.com